CLINICAL TRIAL: NCT07129603
Title: Investigation of the Role of Inflammatory Markers in the Early Detection of Cerebral Vasospasm, Delayed Cerebral Ischemia, and Meningitis Associated With External Cerebrospinal Fluid Drainage After Non-Traumatic Subarachnoid Hemorrhage - A Prospective Case-Control Study
Status: Recruiting | Type: Observational
Sponsor: Tamas Vegh, MD (Other)
Responsible Party: Sponsor-Investigator, Tamas Vegh, MD, MD PhD, University of Debrecen
Organization: University of Debrecen (Other)
Other Study IDs: AITT 2024/3; NNGYK/14357-2/2025 (Other: National Center for Public Health and Pharmacy); DE RKEB/IKEB 6947-2024 (Other: Regional and Institutional Ethics Committee University of Debrecen Clinical Center)
Record Dates: First submitted 2025-08-11; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-04

CONDITIONS: Subarachnoid Haemorrhagic Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background Non-traumatic subarachnoid haemorrhage (SAH) is frequently complicated by delayed cerebral ischaemia (DCI) and by ventriculitis/meningitis when external CSF drains are used; bedside TCCD has limited accuracy for vasospasm detection, creating a need for early biomarkers.

Objective To assess the predictive and diagnostic performance of IL-6, IL-1β, TNFα, procalcitonin (PCT), C-reactive protein (CRP) and adrenomedullin (ADM) measured in CSF and serum for vasospasm, DCI, and drain-associated ventriculitis/meningitis after SAH; to test whether combining biomarkers improves accuracy versus routine parameters; and to explore associations with admission and day-14 serum 25-hydroxy-vitamin D.

Methods Prospective case-control study at the University of Debrecen (planned n≈100; enrolment 01-Nov-2024-31-Dec-2029). Adults with angiography-verified SAH requiring lumbar/ventricular drainage are included; traumatic SAH, prior 6-month meningitis, and immunosuppression are excluded. TCCD is performed daily for 14 days; suspected vasospasm is defined by mean flow velocity >120 cm/s, severe by >200 cm/s, with monitoring extended to day 21 if severe. Sampling: daily CSF IL-6/PCT/CRP until drain removal; IL-1β/TNFα/ADM at 0-2, 3-5, 6-8, 9-11, 12-14 days and at meningitis detection; serum 25-OH-D on drain insertion day and day 14. Outcomes at days 30/90/180: mortality, GOSE, Barthel, Karnofsky, mRS. Statistics: normality testing; t-test or non-parametric equivalents; χ² with Yates' correction; Bonferroni for multiplicity; ROC analysis for diagnostic/predictive performance.

Endpoints DCI: new unexplained CT ischaemia or a new unexplained neurological deficit >1 h. Drain-associated infection: infectologist-adjudicated ventriculitis/meningitis. Vasospasm: TCCD-suggested or DSA-confirmed.

Expected impact An accessible CSF/serum biomarker panel may enable earlier risk stratification and treatment for vasospasm, DCI, and drain-associated infections, and inform future randomized trials of vitamin-D supplementation in SAH.

DETAILED DESCRIPTION:
Brief Summary This single-centre prospective case-control study will evaluate whether a CSF/serum biomarker panel (IL-6, IL-1β, TNFα, PCT, CRP, adrenomedullin) can improve the early diagnosis and risk stratification of cerebral vasospasm, delayed cerebral ischaemia (DCI), and drain-associated ventriculitis/meningitis in adults treated for non-traumatic SAH with external CSF drainage. The study also explores associations with serum 25-hydroxy-vitamin D.

Detailed Description Background: Bedside TCCD is non-invasive but has limited accuracy for vasospasm; DSA is the gold standard but invasive and not easily repeatable. Early, reliable biomarkers could identify high-risk patients sooner. External CSF drainage is standard after SAH but carries a 5-22% risk of ventriculitis/meningitis.

Objectives: Assess diagnostic/predictive performance (including ROC analyses) of IL-6, IL-1β, TNFα, PCT, CRP and adrenomedullin (ADM) in CSF and serum for vasospasm, DCI and drain-associated infection; compare against routine parameters; evaluate combined-biomarker utility; explore associations with 25-OH-vitamin D.

Sampling/monitoring: Daily TCCD for 14 days (extend to day 21 if severe vasospasm); suspected vasospasm if MFV >120 cm/s, severe if >200 cm/s. CSF IL-6/PCT/CRP daily until drain removal; IL-1β, TNFα, ADM at 0-2, 3-5, 6-8, 9-11, 12-14 days and at infection detection; serum 25-OH-vitamin D on drain-insertion day and day 14. Outcomes collected at days 30/90/180 (mortality, GOSE, Barthel, Karnofsky, mRS).

Study Type Observational (Prospective; Case-Control).

Observational Model / Time Perspective Case-Control; Prospective.

Estimated Enrollment

~100 participants.

Outcome Measures Primary Outcome Measures Vasospasm occurrence (binary): TCCD suggestive (MFV >120 cm/s; severe >200 cm/s) and/or DSA-confirmed; diagnostic/predictive performance of biomarkers (e.g., ROC AUC). Time Frame: first 14 days post-ictus (to day 21 if severe vasospasm).

Delayed cerebral ischaemia (DCI) (binary): new unexplained ischaemia on native cranial CT or new unexplained neurological deficit lasting >1 hour; biomarker performance vs DCI status. Time Frame: during acute hospital course (typically within first 14 days).

Drain-associated ventriculitis/meningitis (binary): infectologist-adjudicated diagnosis during drainage; biomarker performance vs infection status. Time Frame: through duration of external drainage.

Secondary Outcome Measures Functional outcomes: mortality; Extended Glasgow Outcome Scale; Barthel Index; Karnofsky; modified Rankin Scale at days 30/90/180 post-ictus.

Comparative accuracy: biomarkers vs routine CSF/blood parameters (e.g., CSF cell count/composition/lactate; albumin & glucose ratios; serum CRP/PCT/IL-6).

Combined-biomarker utility: added value of multi-marker panels over single markers.

Vitamin D exploratory analysis: correlation of biomarkers with admission and day-14 serum 25-OH-vitamin D.

Biospecimen CSF and blood samples collected for biomarker measurements (lab values used for analysis).

Eligibility Criteria

Inclusion:

* Adults (≥18 years).
* Angiography-identifiable non-traumatic SAH (regardless of source).
* Requires lumbar or ventricular drain as part of treatment.

Exclusion:

* Traumatic SAH.
* Patient/legal representative does not consent.
* Meningitis within 6 months prior to ictus.
* Immunosuppressed state (disease or medications affecting WBC number/function).

Groups/Cohorts (for analyses)

* Vasospasm (+/-) (TCCD-suggested or DSA-confirmed vs. absent).
* DCI (+/-) (meets DCI definition vs. absent).
* Drain-associated ventriculitis/meningitis (+/-) (infectologist-adjudicated vs. excluded).

Statistical Plan Normality testing; t-test or non-parametric equivalents; χ² with Yates' correction where appropriate; Bonferroni for multiplicity; ROC analysis for diagnostic/predictive performance.

Location University of Debrecen, Clinical Centre - Department of Anaesthesiology and Intensive Care, Debrecen, Hungary (Neurosurgical Intensive Care Unit).

Contacts Principal Investigator: Prof. Dr. Csilla Molnár - University of Debrecen, Clinical Centre, Department of Anaesthesiology and Intensive Care. (Phone/Email per site policy.)

Keywords Subarachnoid haemorrhage; vasospasm; delayed cerebral ischaemia; ventriculitis; meningitis; IL-6; IL-1β; TNFα; procalcitonin; CRP; adrenomedullin; CSF biomarkers; TCCD; vitamin D.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years).
* Angiography-identifiable non-traumatic SAH (regardless of source).
* Requires lumbar or ventricular drain as part of treatment.

Exclusion Criteria:

* Traumatic SAH.
* Patient/legal representative does not consent.
* Meningitis within 6 months prior to ictus.
* Immunosuppressed state (disease or medications affecting WBC number/function).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (≥18 years) admitted to the Neurosurgical Intensive Care Unit of the University of Debrecen Clinical Centre with non-traumatic subarachnoid haemorrhage (SAH) who, as part of standard care, require external CSF drainage (lumbar or ventricular). Patients are treated per local protocol and monitored with routine severity scales (modified Fisher, Hunt-Hess, WFNS, GCS, VASOGRADE, HAIR). Key exclusions are traumatic SAH, lack of consent, meningitis within the prior 6 months, and clinically relevant immunosuppression. Approximately 100 consecutive eligible patients will be enrolled during the acute hospitalization over the planned inclusion window. The cohort reflects the typical SAH case-mix (both sexes, many critically ill; SAH commonly affects middle-aged adults) and is designed to capture patients at risk for vasospasm, delayed cerebral ischaemia and drain-associated ventriculitis/meningitis under ICU conditions.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
DCI | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Csilla Molnár, MD PhD Full Professor, Principal Investigator — University of Debrecen, Faculty of Medicine, Department of Anaesthesiology and Intensive Care
Locations (1):
- University of Debrecen, Department of Anesthesiology and Intensive Care, Debrecen, Hungary

IPD SHARING:
Plan to Share IPD: Undecided